CLINICAL TRIAL: NCT03194204
Title: Efficacy of Doxycycline as a Combination Therapy in the Treatment of Rheumatoid Arthritis
Brief Title: Re-evaluation of Some Old Rheumatoid Arthritis Therapy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Ibrahem Kamel, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17200080
Record Dates: First submitted 2017-06-10; First posted 2017-06-21 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Doxycycline; Blood Sedimentation; Blood Cell Count; Rheumatoid Factor; epicatechin gallate; C-Reactive Protein; Blood Glucose; Matrix Metalloproteinase 3

STUDY DESIGN:
Intervention Model Description: A group of patients will receive methotrexate only, another group will receive methotrexate plus doxycycline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RA patients treated with methotrexate (Active Comparator): Disease activity score(DAS28) matrix metalloproteinase-3(MMP-3) and matrix metalloproteinase-9(MMP-9), Erythrocyte sedimentation rate C- reactive protein Complete blood count Urine analysis Renal and liver function tests Lipid profile, blood glucose level Serum uric acid Rheumatoid factor (RF IgM, U/L) Anti- cyclic citrullinated peptide . Radiological assessment :Plain radiographs of both hands and feet in the postero-anterior views .
  Cardiac assessment :By electrocardiogram ( ECG ) and echocardiography , Carotid artery intima-medial thickness (IMT) will be done by colored doppler ultrasound.
  Interventions: Drug: Doxycycline Tablets
- RA patients treated with methotrexate plus doxycycline (Active Comparator): Disease activity score(DAS28) Matrix Metalloproteinase-3 (MMP-3) and Matrix Metalloproteinase-9 (MMP-9) Erythrocyte sedimentation rate C- reactive protein Complete blood count Urine analysis Renal and liver function tests Lipid profile, blood glucose level Serum uric acid , Rheumatoid factor (RF IgM(immunoglobulin M), U/L) Anti- cyclic citrullinated peptide. Radiological assessment :Plain radiographs of both hands and feet in the postero-anterior views.
  Cardiac assessment :
  By electrocardiogram ( ECG ) and echocardiography Carotid artery intima-medial thickness (IMT) will be done by colored doppler ultrasound.
  Interventions: Drug: Doxycycline Tablets

INTERVENTIONS:
Drug: Doxycycline Tablets — MMP-3 and MMP-9 will be done with blood samples using ELISA technique CIMT will be done using colored doppler ultrasound
  Other Names: Erythrocyte sedimentation rate (ESR); Complete blood count (CBC).; Lipid profile; Renal and liver function tests; Serum uric acid; Rheumatoid factor (RF IgM, U/L); Anti- cyclic citrullinated peptide; plain radiographs of both hands and feet; electrocardiogram ( ECG ) and echocardiography; Carotid artery intima-medial thickness (CIMT); C-reactive protein (CRP); blood glucose level; Disease activity score(DAS28); Matrix metalloproteinase 3 and 9 (MMP-3)(MMP-9)

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease characterized by joint swelling, joint tenderness and destruction of synovial joints, leading to severe disability and premature mortality.

DETAILED DESCRIPTION:
The rate of cartilage and joint damage in RA is correlated with plasma elevations in inflammatory acute phase reactants, such as C- reactive protein and erythrocyte sedimentation rate, rheumatoid factor positivity and the synovial concentrations of matrix metalloproteinases(MMP), a matrix digesting enzymes directly responsible for joint destruction.

Matrix metalloproteinases (MMP) are a family of zinc-containing endoproteinases that degrade extracellular matrix (ECM) components.The MMPs are thought to play a critical role in the degradation of many components of the extracellular matrix in the synovial joint.

Matrix metalloproteinase-3 (stromelysin-1) is a proteolytic enzyme which is thought to play a pivotal role in joint destruction in RA through breaking down various extracellular components, including collagens (types III, IV, V, IX, and XI), matrix proteins and proteoglycans and activating other pro-MMPs such as pro-MMP-7, pro-MMP-8 and pro-MMP-9.

In RA, MMP-3 is locally produced in the inflamed joint and released into the blood stream. It has been suggested that serum MMP-3 level correlates with levels produced by the synovium, thus reflect the level of activity of rheumatoid synovitis.

MMP-9 has been associated with chronic inflammatory autoimmune diseases. It has been implicated in the pathogenesis of autoimmune diseases.

MMP-9 displays gelatinolytic, elastolytic and collagenolytic activity, thus playing a key role in extracellular matrix turnover, in addition, MMP-9 may also modulate the activity of various biological factors, including other proteinases (e.g., MMP-13), their inhibitors (e.g., α1-antitrypsin) or cytokines.

Matrix metalloproteinases also play key roles in adverse cardiovascular remodeling, atherosclerotic plaque formation and plaque instability, vascular smooth muscle cell (SMC) migration and restenosis that lead to coronary artery disease (CAD) and progressive heart failure.

Matrix metalloproteinases-9 (MMP-9) is mainly found in the most stenotic areas of carotid plaques in humans and is a marker for plaque vulnerability . It can also predict stroke and fatal cardiovascular events . Elevated circulating levels of MMP-9 have been found in subjects with stable angiographic coronary atherosclerosis and intermittent claudication.

The prevalence of athero sclerosis is increased in RA, even in early disease. The earliest vascular change described microscopically in atherosclerosis is intimal media thickening (IMT) , which consists of layers of smooth muscle cells and extracellular matrix. Intimal thickening is more frequent in atherosclerosis-prone arteries such as coronary, carotid, aorta and iliac arteries .

IMT is the "phenotype" of the early phases of atherosclerotic disease and is related to the main traditional risk factors. Moreover, IMT is a marker of organ damage either in the heart or in other vascular districts. The simultaneous measurement of carotid and femoral IMT may improve risk stratification in patients with coronary heart disease.

Atherosclerosis is recognized as a chronic inflammatory condition with key roles for both the innate and adaptive immune systems in the initiation, progression and stability of lesions.

Inflammation is an important trigger of plaque erosion and stability and one focus of secondary prevention of coronary artery disease (CAD) in the general population is the development of anti-inflammatory agents for plaque stabilization.

Many aspects of the pathophysiology of atherosclerosis are mirrored in the inflamed RA synovium, including pronounced infiltration by macro phages and type 1 T-helper cells, collagen degradation and neovascularization . Cytokines such as tumor necrosis factor-α(TNFα), interleukin-6(IL-6) and matrix metalloproteinases are implicated in both processes.

As plaques become more complex, thinning of the fibrous cap occurs. This thinning eventually causes rupture of the plaque, exposing its thrombogenic content to blood, resulting in acute thrombosis and a clinical event .Fibrous cap erosion is thought to be mediated by inflammatory cells, in particular macrophages and T helper cells, via secretion of matrix metalloproteinases.

Doxycycline, a semi-synthetic tetracycline, is a commonly used broad-spectrum antibiotic. It has been shown that it also inhibits the activity of mammalian collagenases and gelatinases, an activity unrelated to its antimicrobial efficacy. Doxycycline not only inhibits MMP-8 and MMP-9 (gelatinase B) activity, but also the synthesis of MMPs in human endothelial cells .

Tetracyclines exhibit multiple anti-inflammatory properties, including the inhibition of T-cell activation and chemotaxis, the downregulation of proinflammatory cytokines, including TNFα and IL-1b and the inhibition of matrixmetalloproteinases.

A study of patients with early disease showed significant efficacy compared with placebo when used in combination with methotrexate .The benefit of minocycline and doxycycline was confirmed in a recent meta-analysis that found clinically significant improvement in disease activity with no increased risk for adverse events. Rheumatologists have not embraced minocycline or doxycycline as primary treatment options for RA and reserve their use primarily in patients with long-standing, refractory disease. Minocycline and doxycycline are safe and moderately effective disease-modifying anti-rheumatic drugs (DMARDs) in the treatment of early rheumatoid arthritis . These drugs are generally well tolerated, with skin complaints, nausea, and dizziness being the most common patient-reported side effects.

Whether RA is caused, triggered, or perpetuated by an infectious agent or agents is still not delineated, it is possible, that suppression of infections in a nonspecific manner, decreasing the stimuli for TNFα production, may play a role in the treatment of RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study are patients with RA (either newly or previously diagnosed) with their age between 18-50 years old having the same normal range of body mass index

Exclusion Criteria:

1. - The investigators will exclude patients with risk factors for atherosclerosis other than rheumatoid arthritis such as:

   * Smoking.
   * Obesity.
   * Hypertension.
   * Diabetes.
   * History of renal or liver diseases.
   * Corticosteroid therapy. 2- Intercurrent infections as they may interfere with levels of metalloproteinases.

     3- Pregnant or lactating females .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
efficacy of doxycycline | 3 months after therapy
  percentage of patients achieving remission or low disease activity as assessed by DAS28
safety of doxycycline in combination with MTX | at day one of the study and every months till the end of the study
  side effects

SECONDARY OUTCOMES:
CIMT as a method for detection of subclinical atherosclerosis in RA patients | 1 day
  colored doppler ultrasound
MMP-3 and 9 as predictors of cardiovascular affection, disease activity and treatment response | day 1 and 3 months follow up
  blood samples using ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdelnaseer M, Elfayomi N, Esmail EH, Kamal MM, Hamdy A, Samie RMA, Elsawy E. Relationship between matrix metalloproteinase-9 and common carotid artery intima media thickness. Neurol Sci. 2016 Jan;37(1):117-122. doi: 10.1007/s10072-015-2358-z. Epub 2015 Aug 30. PMID 26319043
- [Result] Grzela K, Litwiniuk M, Zagorska W, Grzela T. Airway Remodeling in Chronic Obstructive Pulmonary Disease and Asthma: the Role of Matrix Metalloproteinase-9. Arch Immunol Ther Exp (Warsz). 2016 Feb;64(1):47-55. doi: 10.1007/s00005-015-0345-y. Epub 2015 Jun 28. PMID 26123447
- [Result] Ma JD, Zhou JJ, Zheng DH, Chen LF, Mo YQ, Wei XN, Yang LJ, Dai L. Serum matrix metalloproteinase-3 as a noninvasive biomarker of histological synovitis for diagnosis of rheumatoid arthritis. Mediators Inflamm. 2014;2014:179284. doi: 10.1155/2014/179284. Epub 2014 Jul 23. PMID 25147433
- [Result] Mittal B, Mishra A, Srivastava A, Kumar S, Garg N. Matrix metalloproteinases in coronary artery disease. Adv Clin Chem. 2014;64:1-72. doi: 10.1016/b978-0-12-800263-6.00001-x. PMID 24938016
- [Result] Everett BM, Pradhan AD, Solomon DH, Paynter N, Macfadyen J, Zaharris E, Gupta M, Clearfield M, Libby P, Hasan AA, Glynn RJ, Ridker PM. Rationale and design of the Cardiovascular Inflammation Reduction Trial: a test of the inflammatory hypothesis of atherothrombosis. Am Heart J. 2013 Aug;166(2):199-207.e15. doi: 10.1016/j.ahj.2013.03.018. Epub 2013 May 3. PMID 23895801
- [Result] Bernetti M, Abbate R, Cerini G, Gensini GF, Poggesi L, Boddi M. [Carotid and femoral intima-media thickness as an early atherosclerotic marker. Advantages and limits]. G Ital Cardiol (Rome). 2011 Jan;12(1):72-81. Italian. PMID 21428031
- [Result] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Result] Webster G, Del Rosso JQ. Anti-inflammatory activity of tetracyclines. Dermatol Clin. 2007 Apr;25(2):133-5, v. doi: 10.1016/j.det.2007.01.012. PMID 17430750
- [Result] Nakashima Y, Chen YX, Kinukawa N, Sueishi K. Distributions of diffuse intimal thickening in human arteries: preferential expression in atherosclerosis-prone arteries from an early age. Virchows Arch. 2002 Sep;441(3):279-88. doi: 10.1007/s00428-002-0605-1. Epub 2002 Mar 14. PMID 12242525
- [Result] del Rincon ID, Williams K, Stern MP, Freeman GL, Escalante A. High incidence of cardiovascular events in a rheumatoid arthritis cohort not explained by traditional cardiac risk factors. Arthritis Rheum. 2001 Dec;44(12):2737-45. doi: 10.1002/1529-0131(200112)44:123.0.CO;2-%23. PMID 11762933
- [Derived] Ibrahem EM, El-Gendi SS, Mahmoud AA, Abdel-Aal SM, El Nouby FH, El-Deen Mohammed HS. Predictors of Cardiovascular Affection in Patients with Active Rheumatoid Arthritis: Secondary Analysis of a Randomized Controlled Trial. Curr Rheumatol Rev. 2021;17(2):258-266. doi: 10.2174/1573397116666201113090145. PMID 33185166